CLINICAL TRIAL: NCT02887027
Title: Developing an Ecological Momentary Exercise Intervention: Open Trial With Patients
Brief Title: Exercise, Mood and Stress Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Clara Mayo Fellowship (Unknown)
Responsible Party: Principal Investigator, Maria Alexandra Kredlow Acunzo, Graduate Student, Boston University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4017
Record Dates: First submitted 2016-08-07; First posted 2016-09-01 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Anxiety; Post-Traumatic Stress Disorder; Depression
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Group 1 (Experimental): Participants assigned to this group will complete a baseline period of 8 days and an Exercise4Mood Intervention period of 21 days.
  Interventions: Behavioral: Exercise4Mood Intervention
- Exercise Group 2 (Experimental): Participants assigned to this group will complete a baseline period of 11 days and an Exercise4Mood Intervention period of 18 days.
  Interventions: Behavioral: Exercise4Mood Intervention
- Exercise Group 3 (Experimental): Participants assigned to this group will complete a baseline period of 15 days and an Exercise4Mood Intervention period of 14 days.
  Interventions: Behavioral: Exercise4Mood Intervention

INTERVENTIONS:
Behavioral: Exercise4Mood Intervention — The Exercise4Mood Intervention was designed based on principles from the Exercise for Mood and Anxiety protocol (Smits et al., 2009) and consists primarily of a mobile application called Exercise4Mood. It will be supported by text-messages, delivered through SymTrend, reminding participants about their scheduled exercise sessions and prompting them to engage with the app. Its core features include: motivational tips to encourage exercise, reminders about scheduled exercise, tracking of exercise behavior, tracking of mood before, during, and after exercise, and post-exercise positive reinforcement statements.

SUMMARY:
Multiple studies indicate that exercise is effective in treating depressed mood and reducing anxiety sensitivity. As depressive symptoms and anxiety sensitivity are elevated in individuals with anxiety and depressive disorders, exercise could help reduce these symptoms and aid in the overall treatment of these disorders. This project aims to test an ecological momentary exercise intervention (Exercise4Mood) delivered via a mobile phone application in individuals with anxiety or depressive disorders. Previous protocols have tested the acceptability and usability of Exercise4Mood in healthy participants. In Phase 1 of the study, focus groups were conducted to explore the acceptability and usability of the Exercise4Mood app. Qualitative feedback was collected and modifications were made to the app based on this feedback. In Phase 2 of the study, the Exercise4Mood app was tested in 6 healthy participants. Preliminary unpublished findings indicate that the app was acceptable and promoted increased physical activity. The aim of this protocol is to test the acceptability, usability, and efficacy (to improve mood and reduce anxiety) of Exercise4Mood in patients with anxiety or depressive disorders.

DETAILED DESCRIPTION:
Design: A multiple baseline design will be employed: the intervention will be introduced in the 1st participant after a baseline period of 8 days, in the 2nd participant after 11 days, and in the 3rd participant after 15 days. The same pattern will be followed for participants 4-6. Participants will be in the intervention period for 21 days, 18 days, and 14 days respectively, at a prescription of 150 minutes of moderate intensity

Screening Visit:

Individuals who pass the phone screen will be invited to come to our laboratory for remaining screening procedures. At the screening visit, in-person assessment will include informed consent procedures, evaluation of psychiatric inclusion/exclusion criteria and mood, anxiety and traumatic stress disorders with the Anxiety Disorders Interview Schedule for Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 Adult Version (ADIS-5) and additional informal assessment if needed (e.g. to assess eating disorders). The diagnostic assessment will be performed by a study staff member who has been trained in administration of the ADIS-5 and clinical interviewing. If a diagnostic assessment has been conducted at the Center for Anxiety and Related Disorders (CARD) at Boston University within the last six weeks, participants will be given the option to provide consent for it to be used instead (plus additional portions of the ADIS-5 if needed). Eligible participants will be assigned to one of the three conditions above (as this is a single case design, it is not randomized; participants are assigned sequentially to the conditions above). The Screening Visit, which will last 1 hour, may take place on the same or a different day as the pre-baseline visit depending on the researcher and participant's availability.

Pre-Baseline Visit (Day 1):

This in-person visit will occur on Day 1 before the baseline recording period and last 45 minutes. Participants will complete baseline questionnaires and a Physical Activity Recall interview (PAR). Participants' height and weight will be collected. Participants will be given a tutorial on and be provided with an activity and heart monitoring device to wear. Participants will be instructed to engage in their normal level of activity until their next visit. They will be instructed to wear an activity monitor during all waking hours and a heart rate monitor if they exercise. They will be scheduled for a Pre-Intervention Visit either 8, 11, or 15 days later (depending on assignment above).

Pre-Intervention Visit (Day 8, 11, 15 for Participants 1, 2, and 3, respectively):

This in-person visit will occur after the baseline recording period and last 45 minutes. Participants will be prescribed the Exercise4Mood Mobile Intervention for a period 21, 18, or 14 days (depending on assignment above) at a prescription of 150 minutes of moderate intensity (i.e. 64 percent to 76 percent of your maximum heart rate, typically achieved with a brisk walk) exercise per week (as defined by American College of Sports Medicine (ACSM) guidelines).

During this visit, they will complete an introduction to Exercise4Mood. This will involve meeting with the PI who will provide a broad overview of the intervention and training on how to download and use the Exercise4Mood app (and a number to call in case of technical difficulties). Participants will be provided with a Subject ID number and password that they will use to log in to the Exercise4Mood app. They will self-select what days and times they would like to exercise. The PI will help problem solve and ensure that their self-selected plan is feasible. The PI will note down the days and times so that text-message reminders can be sent to the participant. Participants will complete a Physical Activity Recall interview (PAR). Participants will leave the visit with the Exercise4Mood app downloaded on their personal phone and an exercise schedule for the next 21, 18, or 14 days.

Intervention Period (21, 18, or 14 days):

In the two days following the Pre-Intervention Visit, participants will be prompted to complete the Introduction to Exercise4Mood app modules at home. During these modules, they will be provided with information about getting started with exercising. This will include a list of different types of moderate intensity exercise (as listed below) from which participants will self-select what type of exercise they would like to engage in over the intervention period.

* Walking briskly
* Biking slowly
* Jogging
* Swimming leisurely
* Elliptical or other gym machines
* Stair walking
* Basketball
* Aerobic Yoga
* Tennis
* Catch/throw sports (e.g. baseball)

During the intervention period, participants will receive text message prompts to engage with the Exercise4Mood app and engage in exercise. At the end of each week that they are in the intervention, they will be prompted to complete questionnaires through the Exercise4Mood app. These questionnaires will take approximately 15 minutes to complete. During this period, they will wear an activity monitor during all waking hours and a heart rate monitor when they are exercising.

Endpoint Visit (Day 29):

On Day 29, participants will complete an in-person 30 minute visit. During this visit, they will complete an interview about their physical activity engagement, questionnaires (if they did not completed them on the app the day prior), and return the activity and heart rate monitor. Participants will be provided with referrals for mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 to 65.
2. Ability to read and provide informed consent
3. Ownership of an iPhone smartphone device
4. Sedentary as defined as not participating in at least 90 minutes of moderate-intensity exercise per week for at least 3 months.
5. At least minimally active as defined as participating in an average of 10 minutes of mild-intensity physical activity (e.g. walking) per day for the past two weeks.
6. Interest in increasing exercise
7. Daily access to the Internet
8. Current DSM 5 diagnosis of an Anxiety Disorder, Depressive Disorder (i.e. Major Depressive Disorder or Persistent Depressive Disorder), or Post-Traumatic Stress Disorder (PTSD)
9. Sufficient command of the English language

Exclusion Criteria:

1. Participants considered high risk based on the American College Sports Medicine risk stratification guidelines.
2. Participants meeting DSM-5 criteria for a Substance-Related Disorder in the last three months (other than caffeine or nicotine dependence)
3. Participants meeting DSM-5 criteria for past or present Bipolar I or II Disorder or Schizophrenia Spectrum or Other Psychotic Disorder
4. Participants meeting DSM-5 criteria for past or present Eating Disorder
5. Participants endorsing active suicidality, homicidality, or self-destructive acts or urges as assessed through the phone screen and the ADIS
6. Individuals who are not stable (i.e., at the same dosage for at least the past 4 weeks) on psychotropic medications. Current engagement in psychotherapy is permitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Credibility-Expectations Questionnaire (CEQ) | Day 29
  The CEQ is a 6-item self-report questionnaire, which assesses treatment rationale and expectancy. The scale has been used across a number of treatment trials.
Client Satisfaction Questionnaire (CSQ-8) | Day 29
  The CSQ-8 is an 8-item, easily scored and administered measurement that is designed to measure client satisfaction with services. The CSQ-8 is a valid, efficient, and sensitive measure of client satisfaction and has been used across populations and mental health services (Attkisson et al, 1994; Attkisson & Zwick, 1982).
7-Day Physical Activity Recall (PAR) | Change from the start of the baseline period, an expected average of 11 days assessed weekly through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  The is an interviewer-administered procedure assessment of physical activity. Validity and reliability of this technique have been demonstrated (Blair et al., 1985; Sallis et al., 1998) and it has been used in numerous studies. This instrument has been shown to be sensitive to change in studies of moderate intensity activity (Dunn et al., 1998; Dunn et al., 1999).
Physical Activity measured in METS (assessed via Actigraphy) | Change from the start of the baseline period, an expected average of 11 days assessed daily through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  Participants will be lent an ActiGraph (ActiSleep-BT model) wireless activity monitor and Polar heart rate monitor (Polar FT) to wear during the baseline and intervention period. The actigraph is a compact and lightweight device that is worn on an adjustable elastic strap around the waist in conjunction with the heart rate monitor strap that fits securely around the participant's chest area. Participants will be asked to wear the activity monitor during all waking hours and the heart rate monitor only when they are exercising. They will return these devices at the Endpoint Visit.

SECONDARY OUTCOMES:
Anxiety Sensitivity Index (ASI) | Change from the start of the baseline period, an expected average of 11 days assessed weekly through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  The ASI is a 16-item self-report instrument designed to assess one's tendency to respond fearfully to anxiety-related symptoms. The reliability and validity of this measure have been demonstrated (Reiss et al., 1986; Schmidt & Joiner, 2002).
Center for Epidemiological Studies-Depression (CES-D) | Change from the start of the baseline period, an expected average of 11 days assessed weekly through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  The CES-D scale is a short self-report scale designed to measure depressive symptomatology in the general population. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales. The reliability and validity of this measure have been demonstrated (Radloff et al, 1997; Santor et al., 1995).
PTSD Checklist for DSM 5 (PCL) - for individuals with PTSD diagnosis only | Change from the start of the baseline period, an expected average of 11 days assessed weekly through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  The PCL is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD with total scores ranging from 0-80. The PCL is a valid and reliable method of assessing PTSD symptoms in civilian and military populations, across a range of criterion A trauma types (Weathers et al., 2013; Bliese et al., 2008; Harrington & Newman, 2007; Walker et al., 2002).
Depression Anxiety Stress Scale 21 (DASS 21) | Change from the start of the baseline period, an expected average of 11 days assessed weekly through the start of the intervention period, which is expected to last an expected average of 19 days for a total of 30 days
  The DASS 21 is a 21 item self-report questionnaire designed to measure the severity of a range of common symptoms in both depression and anxiety. There are three subscales on the DASS 21 (Depression, Anxiety and Stress) with each subscale score ranging from 0 to 42 and total scores (three subscales added together) ranging from 0 to 126.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Alexandra Kredlow, M.A., Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: Undecided